CLINICAL TRIAL: NCT02820818
Title: Bronchopulmonary Dysplasia: From Neonatal Chronic Lung Disease to Early Onset Adult COPD
Brief Title: Pulmonary Outcomes of Bronchopulmonary Dysplasia in Young Adulthood
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Thuy Mai Luu, Clinical associate professor of pediatrics, St. Justine's Hospital
Other Study IDs: 247649
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Premature Birth; Obstructive Lung Disease; Bronchopulmonary Dysplasia
Keywords: thoracic magnetic resonance imaging; pulmonary function test
MeSH Terms: conditions — Premature Birth; Lung Diseases, Obstructive; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal epithelial cells, whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Preterm birth alters the normal sequence of lung development with lasting respiratory consequences. It is still unclear whether observed respiratory morbidities in preterm born individuals reflect sequelae from a non-progressive lung disease that occurred early in life or result from ongoing active disease that, if left undiagnosed and untreated, could increase the risk of a COPD-like phenotype. We propose to examine micro-structural abnormalities of the lung using innovative non-invasive imaging technologies in relation to pulmonary function and markers of inflammation and oxidative stress in young adults born preterm.

ELIGIBILITY:
Inclusion Criteria:

* 20-29 years old
* For the pre-term subject: <29 weeks gestational age, with or without BPD
* For the matched term control: ≥37 weeks gestational age with birth weight appropriate for gestational age i.e. between the 10th and 90th percentile
* Subject understands the study procedures and is willing to participate in the study as indicated by the signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject is able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater)

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Patient is unable to perform spirometry or plethysmography maneuvers
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants)(at the discretion of the MRI Technologist/3T Manager)
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 25 adults aged 20-29 born preterm (<29 weeks); 25 sex and age-matched controls (friend or sibling).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Lung parenchymal tissue density | Baseline
  Pulmonary hydrogen protons (1H) magnetic resonance imaging (MRI) using ultra-short echo time pulse sequences will be performed to quantify signal intensity (SI) as a surrogate of parenchymal tissue density.

SECONDARY OUTCOMES:
Ventilation defect | Baseline
  Thoracic hyperpolarized 129Xe MRI to measure apparent diffusion coefficient (ADC) - subgroup of 10 participants (5 preterm, 5 control)
Pulmonary function - airflow limitation | Baseline
  Spirometry (FEV1/FVC) will be performed according to the American Thoracic Society guidelines
Pulmonary function - lung volumes | Baseline
  Lung volumes (RV/TLC) by plethysmography will be performed according to the American Thoracic Society guidelines
Pulmonary function - diffusion lung capacity | Baseline
  DLCO will be performed according to the American Thoracic Society guidelines
Pulmonary function - ventilation homogeneity | Baseline
  Lung clearance index by nitrogen washout will be performed according to the American Thoracic Society guidelines

OTHER OUTCOMES:
Inflammatory and oxidative stress markers | Baseline
  Oxidative stress markers glutathione (GSH, GSSG; by capillary zone Electrophoresis) with calculation of Redox potential by the Nernst equation
Pneumoproteins SP-D | Baseline
  Surfactant protein D (plasma)
Pneumoproteins CCSP-16 | Baseline
  CCSP-16 (plasma)

IPD SHARING:
Plan to Share IPD: No